CLINICAL TRIAL: NCT05589857
Title: A Phase II Randomized Controlled Trial to Determine the Efficacy of an auGmented reAlity gaMe in pediatrIc caNcer Patients Who Are Opioid Tolerant Users Undergoing Surgery to Reduce Post-operative Opioid Use
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No Patients Enrolles
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0529; NCI-2022-08945 (Other: NCI- CTRP Clinical Trial Registry)
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Spellbound) (Experimental): Participants will play SpellBound using the iPad's standard camera, which will show you your hospital room and the decal/stickers s as they appear in the real world.
  Interventions: Device: IPAD
- Group 2 (Spellbound) (Experimental): Participants will play the game using augmented reality.
  Interventions: Device: Augmented Reality

INTERVENTIONS:
Device: IPAD — Participants will play a game using the iPad's standard camera, which will show you your hospital room and the decal/stickers s as they appear in the real world.
  Arms: Group 1 (Spellbound)
Device: Augmented Reality — Participants will play a game through (device camera and application) that add virtual or digital characters and items that let participants view the real world.
  Arms: Group 2 (Spellbound)

SUMMARY:
Tto learn if playing an augmented reality game called SpellBound can reduce pain and the need for opioids in young patients following surgery.

DETAILED DESCRIPTION:
Primary Objective:

To assess the efficacy of SpellBound's AR-enabled scavenger hunt to reduce the rate of additional inpatient opioid use in pediatric cancer patients who are chronic/tolerant opioid users undergoing surgery compared to a control non-AR game in a randomized controlled trial.

Secondary Objectives:

To assess the impact of AR versus non-AR control technology in pediatric oncology patients, including:

* Inpatient opioid use
* Average daily inpatient pain score
* Number of opioid requests during hospital stay
* Inpatient PedsQL (quality of life) questionnaire score
* Ambulation/"out of bed" movement
* Number days to discharge-ready status
* Patient experience assessed by satisfaction scores on questionnaire designed by MD Anderson Cancer Center Child Life team
* Outpatient opioid use reported at 30, 60, 90 days.
* Outpatient pain scores reported at 30, 60, 90 days
* Outpatient PedsQL scores reported at 30, 60, and 90 days
* Potential adverse events related to the use of AR (i.e., falls).

ELIGIBILITY:
Inclusion Criteria:

1. Ages 5-15
2. English and Spanish-speaking parents/legal guardians and patients
3. Undergoing surgery requiring postoperative hospitalization is defined as ≥2 hours of duration of surgery and requiring postoperative hospital admission of at least one night
4. Expected to be prescribed postoperative inpatient opioids
5. Prescribed daily opioids for pain for a period equal to or longer than 30 days before surgery.
6. Sufficient cognitive capacity to comprehend and interact with the game. This is defined as the ability to utilize mobile technology (use iPad with or without assistance) and activate and respond to AR experiences within the app as determined by the clinician.
7. Both the child and a legal guardian are willing and able to provide informed consent.

The range from 5-to 15 is based on a recent pilot RCT in which the PI found that older adolescents (>15 years of age) were disinterested in the interactive game.

Exclusion Criteria:

1. Have never taken opioids or have had no daily opioid use within the last 30 days before surgery
2. Inability to demonstrate an understanding of the game from English instructions
3. Any additional concerns based on the study physicians' assessments b. Setting: Academic tertiary cancer center: University of Texas - MD Anderson Cancer Center and Baylor College of Medicine - Texas Children's Hospital

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory | through completion of study, an average of 1 year
  Quality of life assessment: Age-appropriate Pediatric Quality of Life Inventory (PedsQL)29 paper surveys will be administered to the patient (self-report) or guardian (proxy) when patients reach discharge-ready status.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Cata, MD, Principal Investigator — MD Anderson
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT05589857/ICF_000.pdf